CLINICAL TRIAL: NCT05593458
Title: A Multicenter, Randomized, Controlled Study of S-1 Combined With Oxaliplatin by Arterial Infusion Plus PD-1 Antibody Versus Conventional SOX Chemotherapy Plus PD-1 Antibody for Locally Advanced Gastric Cancer
Brief Title: Transarterial Neoadjuvant Chemotherapy vs.Traditional Intravenous Chemotherapy For Locally Advanced Gastric Cancer With SOX+PD-1
Acronym: TACTIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian Chen, Head of Gastrointestinal Surgery, Second affiliated hospital of Zhejiang university School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZEWC_GC_I002
Record Dates: First submitted 2022-10-19; First posted 2022-10-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Gastric Carcinoma
Keywords: gastric cancer; arterial infusion; neoadjuvant therapy; immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arterial infusion group (Experimental): 1. 3 cycles of neoadjuvant chemotherapy: Oxaliplatin arterial infusion+S-1
  2. 3 cycles of immunotherapy: sintilimab
  3. surgery and 3 cycles of adjuvant chemotherapy using SOX regimen plus sintilimab.
  4. S-1 administration till 1 year after surgery
  Interventions: Drug: Oxaliplatin by arterial infusion plus S-1; Drug: Sintilimab neoadjuvant; Procedure: gastrectomy plus D2 lymph node dissection; Drug: SOX adjuvant, Sequential S-1; Drug: Sintilimab adjuvant
- SOX group (Active Comparator): 1. 3 cycles of neoadjuvant chemotherapy: SOX regimen
  2. 3 cycles of immunotherapy: sintilimab
  3. surgery and 3 cycles of adjuvant chemotherapy using SOX regimen plus sintilimab.
  4. S-1 administration till 1 year after surgery
  Interventions: Drug: SOX neoadjuvant; Drug: Sintilimab neoadjuvant; Procedure: gastrectomy plus D2 lymph node dissection; Drug: SOX adjuvant, Sequential S-1; Drug: Sintilimab adjuvant

INTERVENTIONS:
Drug: Oxaliplatin by arterial infusion plus S-1 — 3 cycles oxaliplatin by arterial infusion plus S-1 every 21 days as neoadjuvant chemotherapy.
  Arms: Arterial infusion group
Drug: SOX neoadjuvant — 3 cycles of SOX neoadjuvant chemotherapy every 21 days.
  Arms: SOX group
Drug: Sintilimab neoadjuvant — 3 cycles of neoadjuvant immunotherapy every 21 days.
Procedure: gastrectomy plus D2 lymph node dissection — All patients, whose lesions are resectable and medically operable after 3 cycles neoadjuvant chemotherapy, will receive gastrectomy plus D2 lymph node dissection.
Drug: SOX adjuvant, Sequential S-1 — 3 cycles of SOX adjuvant chemotherapy every 21 days after surgery in both groups.
  Sequential S-1 chemotherapy every 21 days till 1 year postoperation.
Drug: Sintilimab adjuvant — 3 cycles of adjuvant immunotherapy every 21 days.

SUMMARY:
SOX regimen, consisting of oral S-1 and intravenous oxaliplatin, is the preferred regimen for perioperative chemotherapy for gastric cancer. The goal of this clinical trial is to compare the efficacy and safety between S-1 combined with oxaliplatin by arterial infusion, as neoadjuvant chemotherapy, and conventional SOX regimen, in locally advanced gastric cancer. The main question it aims to answer is: whether arterially infused oxaliplatin plus S-1 has the potential to be a better neoadjuvant option for patients with locally advanced gastric cancer.

Participants will be randomised, and receive:

* 3 cycles of conventional SOX chemotherapy plus PD-1 antibody or arterial infused oxaliplatin plus S-1 and PD-1 antibody, as neoadjuvant chemotherapy;
* Adequate gastric resection along with D2 lymph node dissection;
* 3 cycles adjuvant chemotherapy using SOX regimen plus PD-1 antibody.
* Administration of S-1 regularly till 1 year after surgery.

Researchers will compare Major pathological response rate (MPR) ，pathologic complete response rate（pCR）,the 2-year overall survival (OS) rates, 2-year disease free survival (DFS), R0 resection rates, and adverse events, to see if the modified perioperative chemotherapy improve the prognosis of patients with locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group(ECOG) score 0-1
* Ambulatory males or females, aged 18-75 years
* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (Siewert type II or III)
* Locally advanced gastric carcinoma (cT3N2-3M0, cT4aN1-3M0, cT4bNanyM0, American Joint Committee on Cancer (AJCC) TNM staging system 8th edition)
* Life expectancy more than 3 months
* Give written informed consent, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Normal hepatic, renal, and bone marrow function (ALT/AST<2.5 fold of upper limit value;Tbil<1.5mg/dl, Cr<1.5 fold of upper limit value; White Blood Cell count≥3 × 10^9/L, ANC ≥ 1.5 × 10^9/L,PLT≥ 80 × 10^9/L,Hb ≥ 90 g/L).

Exclusion Criteria:

* Patients can not bear surgical procedure.
* Pregnant or lactating women.
* HER2 overexpression(+++) confirmed by immunohistochemistry.
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy.
* History of another malignancy within the last five years.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.
* History of dysphagia, complete or partial gastrointestinal obstruction, active gastrointestinal bleeding and gastrointestinal perforation;
* Organ allografts requiring immunosuppressive therapy.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Moderate or severe renal impairment: serum creatinine > 1.5 x upper limit of normal (ULN).
* Hypersensitivity to any drug of the study regimen.
* With abdominal cavity implantation metastasis or distant metastasis.
* Unwilling or unable to comply with the protocol for the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response rate | 6 months
  The percentage of people who has less than or equal to 10% residual viable tumor after neoadjuvant therapy.

SECONDARY OUTCOMES:
R0 resection rate | 6 months
  The proportion of patients with margin-free resection
2-year Disease Free Rate | 2 years
  The percentage of individuals in this study who are free of the signs and symptoms of gastric cancer at 2 years after treatment
2-year Overall Survival Rate | 2 years
  The percentage of individuals in this study who are alive two years after their diagnosis or the start of treatment.
pathological Complete Response rate | 6 months
  The percentage of people with complete disappearance of all invasive carcinoma cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Department of Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No